CLINICAL TRIAL: NCT01709422
Title: Efficacy and Safety Profiles of Sedation With Propofol Combined With Intravenous Midazolam and Meperidine Versus Intravenous Midazolam and Meperidine for Ambulatory Endoscopic Retrograde-cholangiopancreatography(ERCP).
Brief Title: Efficacy and Safety Profiles of Combination Sedation Propofol With Midazolam and Meperidine.
Acronym: ERCP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Prince of Songkla University (Other)
Responsible Party: Principal Investigator, Nisa Netinatsunton, NKC Institute of Gastroenterology and Hepatology, Prince of Songkla University
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 1774906506805161
Record Dates: First submitted 2012-09-27; First posted 2012-10-18 (Estimated); Results first posted 2013-08-27 (Estimated); Last update posted 2013-10-22 (Estimated); Status verified 2013-09

CONDITIONS: Disorders of Gallbladder, Biliary Tract and Pancrease
Keywords: Propofol; Midazolam; Meperidine
MeSH Terms: interventions — Propofol; Midazolam; Benzodiazepines; Meperidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Propofol (Active Comparator): both midazolam (1mg if aged <= 70 years or 0.5mg in age >70 years) and meperidine 20 mg were given intravenously at the initiation of sedation, Thereafter, an initial bolus of propofol 20 mg intravenously. Sedation was maintained with repeated dose of 5 to 10 mg propofol.
  Interventions: Drug: Propofol; Drug: Midazolam; Drug: Meperidine
- Conventional (Active Comparator): both midazolam 2 to 5 mg and meperidine 25 to 50 mg were given intravenously at the initiation of sedation. Sedation was maintained with repeated doses of 0.5 to 1.0 mg midazolam and 5 to 10 mg meperidine.
  Interventions: Drug: Midazolam; Drug: Meperidine

INTERVENTIONS:
Drug: Propofol — Propofol is the sedative drug used as an additional sedation to one of the study arm.
  Other Names: Diprivan
  Arms: Propofol
Drug: Midazolam — Midazolam is one of the two conventional sedative drugs included in both arms.
  Other Names: Benzodiazepine
Drug: Meperidine — Meperidine is one of the two conventional sedative drugs included in both arms.
  Other Names: Pethidine

SUMMARY:
The purpose of this study is to compare efficacy and safety of combination of propofol and midazolam with meperidine versus midazolam and meperidine for ambulatory ERCP

DETAILED DESCRIPTION:
ERCP is commonly done under sedation with midazolam and meperidine, however some studies showed varying outcomes of this conventional sedation for maintained sedation. Propofol is increasing used for sedation in gastrointestinal procedure owing to its rapid recovery profiles but the complications associated with propofol are not negligible.The investigators prospectively compare the efficacy, induction time, recovery time, patient satisfaction and side effect between propofol based and conventional sedations in patients undergoing ERCP.

ELIGIBILITY:
Inclusion Criteria:

. All outpatients aged more than 18 years who were schedule for ERCP -

Exclusion Criteria:

* pregnant woman
* emergency situation ( i.e. concomitant upper gastrointestinal bleeding, acute cholangitis )
* American Society of Anesthesiologist ( ASA )Class IV or V
* respiratory disease,
* sleep apnea
* allergy to egg or soybean
* drug abuse( benzodiazepine, opioid agonist )
* previous history of failure sedation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2010-06; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nisa Netinatsunton, MD, Principal Investigator — NKC Institute of Gastroenterology and Hepatology, Prince of Songklanakarind University; Nisa Netinatsunton, MD, Principal Investigator — Prince of Songkla University
Locations (1):
- NKC Institues of Gastroenterology and Hepatology, Prince of Songkla University, Hat Yai, Changwat Songkhla, Thailand

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients who were schedule for endoscopic retrograde cholangiopancreatography in NKC Institute ,Prince of Songkla University during January 2010-December 2011
Pre-assignment Details: Patients were excluded from the final analysis if the procedure was terminated due to technical reasons prior to attempted cannulation.
Groups:
- Propofol: The propofol was given as initial bolus of 20 mg and then the dose was given 5-10 mg every 30-60 second.the dose of midazolam was 1 mg in patients below 70 years and 0.5 mg in patients ≥ 70 years and the dose of meperidine was fixed at 20 mg.
- Conventional: The initial dose of midazolam and meperidine were 2-5 mg iv and 25-50 mg iv respectively then the midazolam dose was given 0.5-1.0 mg iv and meperidine dose was given 5-10 mg iv every 2-3 minutes
Period: Overall Study
Arm/Group | Propofol | Conventional
Started | 70 | 70
Completed | 70 | 70
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Propofol,Midazolam and Meperidine: The propofol was given as initial bolus of 20 mg and then the dose was given 5-10 mg every 30-60 second.the dose of midazolam was 1 mg in patients below 70 years and 0.5 mg in patients ≥ 70 years and the dose of meperidine was fixed at 20 mg.
- Midazolam and Meperidine: The initial dose of midazolam and meperidine were 2-5 mg iv and 25-50 mg iv respectively then the midazolam dose was given 0.5-1.0 mg iv and meperidine dose was given 5-10 mg iv every 2-3 minutes
- Total: Total of all reporting groups
Arm/Group | Propofol,Midazolam and Meperidine | Midazolam and Meperidine | Total
Number analyzed (Participants) | 70 | 70 | 140
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 47 | 37 | 84
  >=65 years | 23 | 33 | 56
Age Continuous [Mean (Standard Deviation); unit: years] | 55.77 (17.35) | 61.31 (16.52) | 58.54 (17.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 34 | 72
  Male | 32 | 36 | 68
Region of Enrollment [Number; unit: participants]
  Thailand | 70 | 70 | 140

OUTCOME MEASURES:

1. Secondary Outcome: Cardiovascular Adverse Events.
Description: (1) desaturation(oxygen saturation < 90 % at least 10 second ) (2) hypotension ( systolic blood pressure < 90 mmHg or dropped more than 25 % of baseline ) (3)bradycardia (heart rate < 50 beats/min) and (4) apnea ( cessation of respiratory activity for over 10 seconds ). When patients developed oxygen saturation < 90 %, then nasal oxygen was administered, If patients not able to recover from oxygen therapy and tactile stimulations thus the procedure was terminated. The procedure was terminated if patients developed serious adverse event as heart rate below 5 beats/min and or apnea.
Time Frame: participants will be followed for the duration of procedure, an expected average of 2.0 hours
Population: Intention to treat population include participants who received sedative agents and underwent ERCP.
Measure: Number; unit: Participants
Groups:
- Propofol,Midazolam and Meperidine: the dose of midazolam was 1 mg in patients below 70 years and 0.5 mg in patients ≥ 70 years and the dose of meperidine was fixed at 20 mg. The propofol was given as initial bolus of 20 mg and then the dose was given 5-10 mg every 30-60 second to maintained the desired level of sedation(moderate to deep sedation ) without maximum limit.
- Midazolam and Meperidine: the initial dose of midazolam and meperidine were 2-5 mg iv and 25-50 mg iv respectively then the midazolam dose was given 0.5-1.0 mg iv and meperidine dose was given 5-10 mg iv every 2-3 minutes to maintain the desired level of sedation(moderate to deep sedation ) without maximum limit.
Arm/Group | Propofol,Midazolam and Meperidine | Midazolam and Meperidine
Number analyzed (Participants) | 70 | 70
Participants
  Participants with desatuartion | 26 | 40
  Participants with hypotension | 12 | 14
  Participants with bradycardia | 1 | 0
Statistical Analysis 1: Comparison: Propofol,Midazolam and Meperidine vs Midazolam and Meperidine; Test type: Superiority or Other; p = 0.05, Chi-squared; Risk Difference (RD) = 0.2

2. Primary Outcome: Procedure Related Time
Description: (1) induction time ( the time from sedation to scope intubation ), (2) procedure time ( the time from scope intubation to scope withdrawal ) and (3) recovery time ( the time from scope withdrawal to full recovery ).The induction time, procedural time and recovery time were recorded by the nurse in the endoscopy unit.
Time Frame: participants will be followed for the duration of procedure, an expected average of 2.0 hours ]
Population: Intention to treat population include participants who received sedative agents and underwent endoscopic retrograde cholangiopancreatography(ERCP).
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Propofol,Midazolam and Meperidine: the dose of midazolam was 1 mg in patients below 70 years and 0.5 mg in patients ≥ 70 years and the dose of meperidine was fixed at 20 mg. The propofol was given as initial bolus of 20 mg and then the dose was given 5-10 mg every 30-60 second to maintained the desired level of sedation (moderate to deep sedation ) without maximum limit
- Midazolam and Meperidine: the initial dose of midazolam and meperidine were 2-5 mg iv and 25-50 mg iv respectively then the midazolam dose was given 0.5-1.0 mg iv and meperidine dose was given 5-10 mg iv every 2-3minutes to maintain the desired level of sedation (moderate to deep sedation ) without maximum limit.
Arm/Group | Propofol,Midazolam and Meperidine | Midazolam and Meperidine
Number analyzed (Participants) | 70 | 70
minutes
  procedure time | 40.67 (27.50) | 43.24 (31.35)
  induction time | 3.94 (2.18) | 5.47 (2.51)
  recovery time | 24.71 (23.03) | 88.50 (54.62)
Statistical Analysis 1: Comparison: Propofol,Midazolam and Meperidine vs Midazolam and Meperidine; Test type: Superiority or Other; p = 0.05, t-test, 2 sided; Mean Difference (Final Values) = 28

ADVERSE EVENTS:
Time Frame: 1 month
Description: ERCP complications and sedation related complications are assessed one month after the procedure date.
Arm/Group | Propofol,Midazolam and Meperidine | Midazolam and Meperidine
Serious Adverse Events (participants affected / at risk) | 1/70 | 0/70
Other Adverse Events (participants affected / at risk) | 26/70 | 40/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Propofol,Midazolam and Meperidine (N=70) | Midazolam and Meperidine (N=70)
Severe bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Propofol,Midazolam and Meperidine (N=70) | Midazolam and Meperidine (N=70)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 26 (26) | 40 (40)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No